CLINICAL TRIAL: NCT02833142
Title: A Randomized, Blinded, Parallel-Group, Phase 1 Study of Pharmacokinetics, Safety and Tolerability of Single Intravenous Doses of BIIB033 (Opicinumab ) Produced by 2 Manufacturing Processes, in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety and Tolerability of Single Doses of BIIB033 (Opicinumab) Produced by 2 Manufacturing Processes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 215HV103
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis; Acute Optic Neuritis
Keywords: Healthy Volunteer; opicinumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIIB033-A (Experimental): Staggered single dosing schema
  Interventions: Drug: BIIB033 (opicinumab)
- BIIB033-B (Experimental): Staggered single dosing schema
  Interventions: Drug: BIIB033 (opicinumab)

INTERVENTIONS:
Drug: BIIB033 (opicinumab)

SUMMARY:
The primary objective of the study is to characterize the pharmacokinetics (PK) of BIIB033-B and to compare the PK profile with that of BIIB033-A in healthy volunteers. Secondary objectives are: To assess the safety and tolerability of BIIB033-A and BIIB033-B; To assess the secondary PK parameters of BIIB033-A and BIIB033-B; To assess the immunogenicity of BIIB033-A and BIIB033-B.

ELIGIBILITY:
Key Inclusion Criteria:

* - Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
* - Must have a body mass index of 18 to 32 kg/m2, inclusive.
* - All male participants and all female participants of childbearing potential must practice highly effective methods of contraception during the study and be willing and able to continue contraception for 6 months after being dosed with study treatment. Male participants must not have unprotected sexual intercourse with a female who is pregnant or breastfeeding during the study. Male participants must also be willing to refrain from sperm donation for at least 6 months after dosing with study treatment.
* - Must be in good health as determined by the Investigator (or designee), based on medical history and screening evaluations.

Key Exclusion Criteria:

* - History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal or other major disease, as determined by the Investigator.
* - History of or ongoing malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 12 months prior to Day -1).
* - Serious infection (e.g., pneumonia, septicemia) as determined by the Investigator, within the 3 months prior to Day -1.
* - Fever or bacterial or viral infection (including upper respiratory tract infection) within 2 weeks prior to Day -1.
* - History of severe allergic or anaphylactic reactions, or history of any allergic reaction that in the opinion of the Investigator is likely to be exacerbated by any component of the study treatment.
* - Prior exposure to BIIB033.
* - Female participants who are breastfeeding or pregnant at Screening or Day -1, or plan to become pregnant during the study or during the 6 months following study drug administration.
* - History of, or positive test result at Screening for, human immunodeficiency virus.
* - History of, or positive test result at Screening for, hepatitis C virus antibody or hepatitis B virus (defined as positive for hepatitis B surface antigen or hepatitis B core antibody).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PK parameter of BIIB033: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Up to Day 89
PK parameter of BIIB033: Area under the concentration-time curve from time 0 to Day 85 (AUC84d) | Day 85
PK parameter of BIIB033: Maximum observed concentration (Cmax) | Up to Day 89

SECONDARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 17 weeks
Number of participants with clinically significant laboratory parameters | Up to 17 weeks
Number of participants with clinically significant vital sign abnormalities | Up to 17 weeks
Number of participants with clinically significant electrocardiograms (ECGs) abnormalities | Up to 17 weeks
Number of participants with clinically significant physical examination abnormalities | Up to 17 weeks
PK parameter of BIIB033: Time to reach maximum observed concentration (Tmax) | Up to Day 89
PK parameter of BIIB033: Terminal elimination half-life (t1/2) | Up to Day 89
PK parameter of BIIB033: Volume of distribution at steady state (Vss) | Up to Day 89
PK parameter of BIIB033: Clearance (CL) | Up to Day 89
Number of participants with presence of anti-BIIB033 antibodies | Pre-dose, Day 22 and Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Madison, Wisconsin, United States